CLINICAL TRIAL: NCT03611257
Title: Effect of Direct Rapid Antibiotic Susceptibility Testing (dRAST) on Treatment for Bacteremia in Patients With Hematologic Diseases: Randomized Controlled Trial
Brief Title: Effect of dRAST on Treatment for Bacteremia in Patients With Hematologic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wan Beom Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1806-173-955
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Hematologic Diseases; Bacteremia Sepsis
Keywords: Bacteremia; Optimal targeted antibiotics; Antibiotic susceptibility test; Antimicrobial stewardship
MeSH Terms: conditions — Hematologic Diseases; Bacteremia

STUDY DESIGN:
Intervention Model Description: Single center prospective randomised clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dRAST (Experimental): Hematologic patients with bacteremia will receive antibiotics based on "dRAST" results.
  Interventions: Diagnostic Test: dRAST
- Current standard method (Active Comparator): Hematologic patients with bacteremia will receive antibiotics based on current standard method results.
  Interventions: Diagnostic Test: Current standard method

INTERVENTIONS:
Diagnostic Test: dRAST — Infectious diseases specialists will do active antimicrobial stewardship according to dRAST results in addition to Gram staining results and current standard method.
  Arms: dRAST
Diagnostic Test: Current standard method — Infectious diseases specialists will do active antimicrobial stewardship according to Gram staining results, and current standard method without dRAST results.
  Arms: Current standard method

SUMMARY:
The purpose of this study is to evaluate whether the use of direct rapid antibiotic susceptibility test (dRAST), in addition to the current standard antibiotic susceptibility test, can increase the proportion of patients with hematologic disease who received appropriate antibiotics in early period of bacteremia.

DETAILED DESCRIPTION:
* patients with hematologic diseases who have high risk of bacteremia, because of immune suppression treatment or intensive chemotherapy or bone marrow transplantation which these patients had received, will be recruited in tertiary referral medical centers.
* All the participants will be randomly assigned into either dRAST group or current standard antibiotic susceptibility test group.
* All the participants in the both arms will receive antimicrobial stewardship by infectious disease specialists. Antimicrobial stewardship will be performed at each timepoint of Gram stain results reporting, dRAST results reporting, and current method reporting.
* Target numbers are 58 and 58, respectively.
* All the participants will be monitored for general medical conditions such as vital sign and response to antibiotic treatment by infectious disease specialists for 1 week.
* The percentage of patients who received optimal targeted antibiotics 72 hours after blood collection for blood culture will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are expected to be admitted for more than 2 days due to treatment or complications of hematologic diseases (acute leukemia, chronic leukemia, myelodysplastic syndrome, lymphoma, multiple myeloma, aplastic anemia, etc.) in Seoul National University Hospital.
* Patients with confirmed bacteremia
* Patients who can understand the details of the clinical trial's explanation and provide the written consent

Exclusion Criteria:

* Patients who are expected to stay in the hospital within 2 days
* Patients without bacteremia during hospitalization
* Patients who show fungemia without evidence of bacteremia

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients receiving optimal targeted antibiotics 72 hours after blood collection for blood culture | 72 hour after blood culture collection
  The percentage of patients receiving optimal targeted antibiotics antibiotics which is defined as most effective and narrowest antibiotics based on susceptibility testing results, 72 hours after blood collection for blood culture

SECONDARY OUTCOMES:
Time to optimal targeted antibiotics | Time from first blood culture collection up to 1 month
  The time to the optimal targeted antibiotics administration after blood culture collection
Amount of broad-spectrum antibiotics use | Time from first blood culture collection up to 1 week
  The duration of use of major antibiotics (vancomycin, carbapenem)
Time to defervescence | Time from first blood culture collection up to 1 month
  Time from the time of blood culture collection to the time of fever resolution
proportion of positive blood culture 48 hours after first blood culture | Time from blood culture collection up to 1 month
  proportion of positive blood culture 48 hours after first blood culture
30-day mortality rate related with bacteremia | Time from blood culture collection up to 30-day
  30-day mortality rate related with bacteremia
Percentage of patients receiving optimal targeted antibiotics 48 hours after | 48 hour after blood culture collection
  The percentage of patients receiving optimal targeted antibiotics antibiotics which is defined as most effective and narrowest antibiotics based on susceptibility testing results, 48 hours after blood collection for blood culture
Percentage of patients receiving unnecessary broad spectrum antibiotics 48 hours after | 48 hour after blood culture collection
  The percentage of patients receiving unnecessary broad spectrum antibiotics which is defined as administration of antibiotics to which organisms were susceptible, but had broad-spectrum activity requiring de-escalation or discontinuing administration, 48 hours after blood collection for blood culture
Percentage of patients receiving unnecessary broad spectrum antibiotics 72 hours after | 72 hour after blood culture collection
  The percentage of patients receiving unnecessary broad spectrum antibiotics which is defined as administration of antibiotics to which organisms were susceptible, but had broad-spectrum activity requiring de-escalation or discontinuing administration, 72 hours after blood collection for blood culture
Percentage of patients receiving ineffective antibiotics 48 hours after | 48 hour after blood culture collection
  The percentage of patients receiving ineffective antibiotics which is defined if the organisms were not susceptible, 48 hours after blood collection for blood culture
Percentage of patients receiving ineffective antibiotics 72 hours after | 72 hour after blood culture collection
  The percentage of patients receiving ineffective antibiotics which is defined if the organisms were not susceptible, 72 hours after blood collection for blood culture

CONTACTS AND LOCATIONS:
Overall Officials: wbpark1@snu.ac.kr Park, M.D., PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
We are not planning to share IPDs publically, but de-identified individual participant data for all outcome measures could be shared with other researchers under their request.

REFERENCES:
- [Background] Choi J, Yoo J, Lee M, Kim EG, Lee JS, Lee S, Joo S, Song SH, Kim EC, Lee JC, Kim HC, Jung YG, Kwon S. A rapid antimicrobial susceptibility test based on single-cell morphological analysis. Sci Transl Med. 2014 Dec 17;6(267):267ra174. doi: 10.1126/scitranslmed.3009650. PMID 25520395
- [Background] Choi J, Jeong HY, Lee GY, Han S, Han S, Jin B, Lim T, Kim S, Kim DY, Kim HC, Kim EC, Song SH, Kim TS, Kwon S. Direct, rapid antimicrobial susceptibility test from positive blood cultures based on microscopic imaging analysis. Sci Rep. 2017 Apr 25;7(1):1148. doi: 10.1038/s41598-017-01278-2. PMID 28442767
- [Background] Huh HJ, Song DJ, Shim HJ, Kwon WK, Park MS, Ryu MR, Cho EH, Oh J, Yoo IY, Lee NY. Performance evaluation of the QMAC-dRAST for staphylococci and enterococci isolated from blood culture: a comparative study of performance with the VITEK-2 system. J Antimicrob Chemother. 2018 May 1;73(5):1267-1271. doi: 10.1093/jac/dky015. PMID 29415214
- [Background] Kumar A, Roberts D, Wood KE, Light B, Parrillo JE, Sharma S, Suppes R, Feinstein D, Zanotti S, Taiberg L, Gurka D, Kumar A, Cheang M. Duration of hypotension before initiation of effective antimicrobial therapy is the critical determinant of survival in human septic shock. Crit Care Med. 2006 Jun;34(6):1589-96. doi: 10.1097/01.CCM.0000217961.75225.E9. PMID 16625125
- [Background] Garnacho-Montero J, Aldabo-Pallas T, Garnacho-Montero C, Cayuela A, Jimenez R, Barroso S, Ortiz-Leyba C. Timing of adequate antibiotic therapy is a greater determinant of outcome than are TNF and IL-10 polymorphisms in patients with sepsis. Crit Care. 2006;10(4):R111. doi: 10.1186/cc4995. PMID 16859504
- [Background] Bauer KA, Perez KK, Forrest GN, Goff DA. Review of rapid diagnostic tests used by antimicrobial stewardship programs. Clin Infect Dis. 2014 Oct 15;59 Suppl 3:S134-45. doi: 10.1093/cid/ciu547. PMID 25261540
- [Background] Renders NH, Kluytmans JA, Verbrugh HA. Clinical impact of rapid in vitro susceptibility testing and bacterial identification. J Clin Microbiol. 1995 Feb;33(2):508. doi: 10.1128/jcm.33.2.508-508.1995. No abstract available. PMID 7714220
- [Background] Klastersky J, Ameye L, Maertens J, Georgala A, Muanza F, Aoun M, Ferrant A, Rapoport B, Rolston K, Paesmans M. Bacteraemia in febrile neutropenic cancer patients. Int J Antimicrob Agents. 2007 Nov;30 Suppl 1:S51-9. doi: 10.1016/j.ijantimicag.2007.06.012. Epub 2007 Aug 8. PMID 17689933